CLINICAL TRIAL: NCT00012558
Title: Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: N01MH80001 (NIH); DSIR AT
Record Dates: First submitted 2001-03-13; First posted 2001-03-15 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-04

CONDITIONS: Bipolar Disorder
Keywords: Psychotic Disorders; Mood Disorders; Manic-Depressive Illness; Hypomania; Mania; Mood Stabilizer
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Mood Disorders; Major Affective Disorder 2; Mania | interventions — Lithium; Valproic Acid; Bupropion; Paroxetine; Lamotrigine; Risperidone; Inositol; Tranylcypromine; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: lithium
Drug: valproate
Drug: bupropion
Drug: paroxetine
Drug: lamotrigine
Drug: risperidone
Drug: inositol
Drug: tranylcypromine
Behavioral: Cognitive Behavioral Therapy
Behavioral: Family-focused Therapy
Behavioral: Interpersonal and Social Rhythms Therapy

SUMMARY:
A long-term study of current treatments for bipolar disorder, including medications and psychosocial therapies.

DETAILED DESCRIPTION:
STEP-BD is evaluating all the best-practice treatment options used for bipolar disorder: mood-stabilizing medications, antidepressants, atypical antipsychotics, and psychosocial interventions - or "talk" therapies - including Cognitive Behavioral Therapy, Family-focused Therapy, Interpersonal and Social Rhythm Therapy, and Collaborative Care (psychoeducation).

There are two kinds of treatment "pathways" in STEP-BD, and participants may have the opportunity to take part in both. The medications and psychosocial interventions provided in these pathways are considered among the best choices of treatment for bipolar disorder in everyday clinical practice.

In the "Best Practice Pathway," participants are followed by a STEP-BD certified doctor and all treatment choices are individualized. Everyone enrolled in STEP-BD may participate in this pathway. Participants and their doctors work together to decide on the best treatment plans and to change these plans if needed. Also, anyone who wishes to stay on his or her current treatment upon entering STEP-BD may do so in this pathway. Adolescents and adults age 15 years and older may participate in the Best Practice Pathway.

For adults age 18 and older, another way to participate is in the STEP-BD "Randomized Care Pathways." Depending on their symptoms, participants may be offered treatment in one or more of these pathways during the course of the study. The participants remain on mood-stabilizing medication. However, because doctors are uncertain which of several treatment strategies work best for bipolar disorder, another medication and/or talk therapy may be added. Each Randomized Care Pathway involves a different set of these additional treatments.

Unlike in the Best Practice Pathway, the participants in the Randomized Care Pathways are randomly assigned to treatments. Also, in some cases, neither the participant nor the doctor will be told which of the different medications is being added. This is called a "double-blind" study and is done so that the medication effects can be evaluated objectively, without any unintended bias that may come from knowing what has been assigned. Participants will not be assigned medications that they have had bad reactions to in the past, that they are strongly opposed to, or that the doctor feels are unsuitable for them. The medication(s) participants may be randomly assigned to in the Randomized Care Pathways are free of charge. There are other treatment options for participants if they do not respond well to the treatment assigned to them. Also, participants may return to the Best Practice Pathway at any time. About 1,500 individuals will be enrolled in at least one Randomized Care Pathway during their period of participation in STEP-BD.

It is important to note that STEP-BD provides continuity of care. For example, if a participant starts out in the Best Practice Pathway and later chooses to enter one of the Randomized Care Pathways, he or she continues with the same STEP-BD doctor and treatment team. Then, after completing the Randomized Care Pathway, the participant may return to the Best Practice Pathway for ongoing, individually-tailored treatment.

ELIGIBILITY:
General Inclusion Criteria:

* current age 15 or older (Best Practice Pathway) or 18 years or older (Randomized Care Pathways);
* able to give informed consent for data to be harvested;
* meet DSM-IV criteria for Bipolar I Disorder, Bipolar II Disorder, Bipolar Disorder NOS, or Cyclothymic Disorder;
* undergo a complete standard evaluation including clinical interview, self ratings, and laboratory studies;
* meet with Clinical Specialist as scheduled;
* able to complete all Study Registry Forms within 3 months of registration.

General Exclusion Criteria:

* unwilling or unable to adhere to basic study requirements (i.e., complete rating forms, or attend scheduled evaluations);
* not competent to give informed consent in the opinion of the investigator (e.g., psychotic).

Participants will be asked to remain in the study for up to five years so that the investigators can document and evaluate long-term treatment outcome. Participants will meet with their STEP-BD psychiatrist for periodic evaluations and/or treatment adjustments during the course of the study, fill out various self-rating forms, and when applicable, participate in psychotherapy. One of the psychotherapy options, Family-Focused Therapy, will require participants and their families to attend counseling sessions together. Overall, the estimated amount of time required from participants in the study is 2 to 4 hours per month.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000
Dates: Start 1998-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Gary Sachs, M.D., Principal Investigator — Massachusetts General Hospital; Michael Thase, M.D., Principal Investigator — University of Pittsburgh
Locations (11):
- United States (11):
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado, Colorado Psychiatric Health Clinical Investigation Center, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Tulsa, Oklahoma
  - Portland Veteran's Administration Medical Center, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Sachs GS, Thase ME, Otto MW, Bauer M, Miklowitz D, Wisniewski SR, Lavori P, Lebowitz B, Rudorfer M, Frank E, Nierenberg AA, Fava M, Bowden C, Ketter T, Marangell L, Calabrese J, Kupfer D, Rosenbaum JF. Rationale, design, and methods of the systematic treatment enhancement program for bipolar disorder (STEP-BD). Biol Psychiatry. 2003 Jun 1;53(11):1028-42. doi: 10.1016/s0006-3223(03)00165-3. PMID 12788248
- [Background] Sachs GS, Guille C, McMurrich SL. A clinical monitoring form for mood disorders. Bipolar Disord. 2002 Oct;4(5):323-7. doi: 10.1034/j.1399-5618.2002.01195.x. PMID 12479665
- [Background] Sachs GS. Strategies for improving treatment of bipolar disorder: integration of measurement and management. Acta Psychiatr Scand Suppl. 2004;(422):7-17. doi: 10.1111/j.1600-0447.2004.00409.x. PMID 15330934
- [Background] Thase ME, Bhargava M, Sachs GS. Treatment of bipolar depression: current status, continued challenges, and the STEP-BD approach. Psychiatr Clin North Am. 2003 Jun;26(2):495-518. doi: 10.1016/s0193-953x(03)00029-7. PMID 12778844
- [Background] Perlick DA, Wolff N, Miklowitz DJ, Menard K, Rosenheck RR, & STEP-BD Family Experience Collaborative Study Group [abstract]. Development of an Integrated Model of Family Burden in Bipolar Illness. The Journal of Mental Health Policy and Economics 6(Supplemental): 37, 2003.
- [Background] Gray SM, Frankle WG, Sachs GS. STEP BD: A design for evaluating effectiveness of treatment for bipolar disorder. The Economics of Neuroscience 3(1): 65-68, 2001.
- [Result] Lembke A, Miklowitz DJ, Otto MW, Zhang H, Wisniewski SR, Sachs GS, Thase ME, Ketter TA; STEP-BD Investigators. Psychosocial service utilization by patients with bipolar disorders: data from the first 500 participants in the Systematic Treatment Enhancement Program. J Psychiatr Pract. 2004 Mar;10(2):81-7. doi: 10.1097/00131746-200403000-00002. PMID 15330403
- [Result] Perlis RH, Miyahara S, Marangell LB, Wisniewski SR, Ostacher M, DelBello MP, Bowden CL, Sachs GS, Nierenberg AA; STEP-BD Investigators. Long-term implications of early onset in bipolar disorder: data from the first 1000 participants in the systematic treatment enhancement program for bipolar disorder (STEP-BD). Biol Psychiatry. 2004 May 1;55(9):875-81. doi: 10.1016/j.biopsych.2004.01.022. PMID 15110730
- [Result] Simon NM, Otto MW, Weiss RD, Bauer MS, Miyahara S, Wisniewski SR, Thase ME, Kogan J, Frank E, Nierenberg AA, Calabrese JR, Sachs GS, Pollack MH; STEP-BD Investigators. Pharmacotherapy for bipolar disorder and comorbid conditions: baseline data from STEP-BD. J Clin Psychopharmacol. 2004 Oct;24(5):512-20. doi: 10.1097/01.jcp.0000138772.40515.70. PMID 15349007
- [Result] Marangell LB, Martinez JM, Ketter TA, Bowden CL, Goldberg JF, Calabrese JR, Miyahara S, Miklowitz DJ, Sachs GS, Thase ME; STEP-BD Investigators. Lamotrigine treatment of bipolar disorder: data from the first 500 patients in STEP-BD. Bipolar Disord. 2004 Apr;6(2):139-43. doi: 10.1111/j.1399-5618.2004.00098.x. PMID 15005752
- [Result] Schneck CD, Miklowitz DJ, Calabrese JR, Allen MH, Thomas MR, Wisniewski SR, Miyahara S, Shelton MD, Ketter TA, Goldberg JF, Bowden CL, Sachs GS. Phenomenology of rapid-cycling bipolar disorder: data from the first 500 participants in the Systematic Treatment Enhancement Program. Am J Psychiatry. 2004 Oct;161(10):1902-8. doi: 10.1176/ajp.161.10.1902. PMID 15465989
- [Result] Kogan JN, Otto MW, Bauer MS, Dennehy EB, Miklowitz DJ, Zhang HW, Ketter T, Rudorfer MV, Wisniewski SR, Thase ME, Calabrese J, Sachs GS; STEP-BD Investigators. Demographic and diagnostic characteristics of the first 1000 patients enrolled in the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). Bipolar Disord. 2004 Dec;6(6):460-9. doi: 10.1111/j.1399-5618.2004.00158.x. PMID 15541061
- [Result] Simon NM, Otto MW, Wisniewski SR, Fossey M, Sagduyu K, Frank E, Sachs GS, Nierenberg AA, Thase ME, Pollack MH. Anxiety disorder comorbidity in bipolar disorder patients: data from the first 500 participants in the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). Am J Psychiatry. 2004 Dec;161(12):2222-9. doi: 10.1176/appi.ajp.161.12.2222. PMID 15569893
- [Result] Morris CD, Miklowitz DJ, Wisniewski SR, Giese AA, Thomas MR, Allen MH. Care satisfaction, hope, and life functioning among adults with bipolar disorder: data from the first 1000 participants in the Systematic Treatment Enhancement Program. Compr Psychiatry. 2005 Mar-Apr;46(2):98-104. doi: 10.1016/j.comppsych.2004.07.026. PMID 15723025
- [Result] Allen MH, Chessick CA. Instability of symptoms in recurrent major depression. Am J Psychiatry. 2005 Feb;162(2):403; author reply 403-4. doi: 10.1176/appi.ajp.162.2.403. No abstract available. PMID 15677618
- [Result] Nierenberg AA, Miyahara S, Spencer T, Wisniewski SR, Otto MW, Simon N, Pollack MH, Ostacher MJ, Yan L, Siegel R, Sachs GS; STEP-BD Investigators. Clinical and diagnostic implications of lifetime attention-deficit/hyperactivity disorder comorbidity in adults with bipolar disorder: data from the first 1000 STEP-BD participants. Biol Psychiatry. 2005 Jun 1;57(11):1467-73. doi: 10.1016/j.biopsych.2005.01.036. PMID 15950022
- [Result] Weiss RD, Ostacher MJ, Otto MW, Calabrese JR, Fossey M, Wisniewski SR, Bowden CL, Nierenberg AA, Pollack MH, Salloum IM, Simon NM, Thase ME, Sachs GS; for STEP-BD Investigators. Does recovery from substance use disorder matter in patients with bipolar disorder? J Clin Psychiatry. 2005 Jun;66(6):730-5; quiz 808-9. doi: 10.4088/jcp.v66n0609. PMID 15960566
- [Result] Fagiolini A, Kupfer DJ, Masalehdan A, Scott JA, Houck PR, Frank E. Functional impairment in the remission phase of bipolar disorder. Bipolar Disord. 2005 Jun;7(3):281-5. doi: 10.1111/j.1399-5618.2005.00207.x. PMID 15898966
- [Result] Nierenberg AA, Ostacher MJ, Calabrese JR, Ketter TA, Marangell LB, Miklowitz DJ, Miyahara S, Bauer MS, Thase ME, Wisniewski SR, Sachs GS. Treatment-resistant bipolar depression: a STEP-BD equipoise randomized effectiveness trial of antidepressant augmentation with lamotrigine, inositol, or risperidone. Am J Psychiatry. 2006 Feb;163(2):210-6. doi: 10.1176/appi.ajp.163.2.210. PMID 16449473
- [Result] Perlis RH, Ostacher MJ, Patel JK, Marangell LB, Zhang H, Wisniewski SR, Ketter TA, Miklowitz DJ, Otto MW, Gyulai L, Reilly-Harrington NA, Nierenberg AA, Sachs GS, Thase ME. Predictors of recurrence in bipolar disorder: primary outcomes from the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). Am J Psychiatry. 2006 Feb;163(2):217-24. doi: 10.1176/appi.ajp.163.2.217. PMID 16449474
- [Result] Fossey MD, Otto MW, Yates WR, Wisniewski SR, Gyulai L, Allen MH, Miklowitz DJ, Coon KA, Ostacher MJ, Neel JL, Thase ME, Sachs GS, Weiss RD; Step-BD Investigators. Validity of the distinction between primary and secondary substance use disorder in patients with bipolar disorder: data from the first 1000 STEP-BD participants. Am J Addict. 2006 Mar-Apr;15(2):138-43. doi: 10.1080/10550490500528423. PMID 16595351
- [Result] Zhang H, Wisniewski SR, Bauer MS, Sachs GS, Thase ME; Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) Investigators. Comparisons of perceived quality of life across clinical states in bipolar disorder: data from the first 2000 Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) participants. Compr Psychiatry. 2006 May-Jun;47(3):161-8. doi: 10.1016/j.comppsych.2005.08.001. PMID 16635643
- [Result] Joffe H, Kim DR, Foris JM, Baldassano CF, Gyulai L, Hwang CH, McLaughlin WL, Sachs GS, Thase ME, Harlow BL, Cohen LS. Menstrual dysfunction prior to onset of psychiatric illness is reported more commonly by women with bipolar disorder than by women with unipolar depression and healthy controls. J Clin Psychiatry. 2006 Feb;67(2):297-304. doi: 10.4088/jcp.v67n0218. PMID 16566627
- [Result] Joffe H, Cohen LS, Suppes T, McLaughlin WL, Lavori P, Adams JM, Hwang CH, Hall JE, Sachs GS. Valproate is associated with new-onset oligoamenorrhea with hyperandrogenism in women with bipolar disorder. Biol Psychiatry. 2006 Jun 1;59(11):1078-86. doi: 10.1016/j.biopsych.2005.10.017. Epub 2006 Jan 31. PMID 16448626
- [Result] Sachs GS, Yan LJ, Swann AC, Allen MH. Integration of suicide prevention into outpatient management of bipolar disorder. J Clin Psychiatry. 2001;62 Suppl 25:3-11. PMID 11765093
- [Result] Waxmonsky JA, Thomas MR, Miklowitz DJ, Allen MH, Wisniewski SR, Zhang H, Ostacher MJ, Fossey MD. Prevalence and correlates of tobacco use in bipolar disorder: data from the first 2000 participants in the Systematic Treatment Enhancement Program. Gen Hosp Psychiatry. 2005 Sep-Oct;27(5):321-8. doi: 10.1016/j.genhosppsych.2005.05.003. PMID 16168792
- [Result] Martinez JM, Marangell LB, Simon NM, Miyahara S, Wisniewski SR, Harrington J, Pollack MH, Sachs GS, Thase ME. Baseline predictors of serious adverse events at one year among patients with bipolar disorder in STEP-BD. Psychiatr Serv. 2005 Dec;56(12):1541-8. doi: 10.1176/appi.ps.56.12.1541. PMID 16339616
- [Result] Goldberg JF, Allen MH, Miklowitz DA, Bowden CL, Endick CJ, Chessick CA, Wisniewski SR, Miyahara S, Sagduyu K, Thase ME, Calabrese JR, Sachs GS. Suicidal ideation and pharmacotherapy among STEP-BD patients. Psychiatr Serv. 2005 Dec;56(12):1534-40. doi: 10.1176/appi.ps.56.12.1534. PMID 16339615
- [Result] Allen MH, Chessick CA, Miklowitz DJ, Goldberg JF, Wisniewski SR, Miyahara S, Calabrese JR, Marangell L, Bauer MS, Thomas MR, Bowden CL, Sachs GS. Contributors to suicidal ideation among bipolar patients with and without a history of suicide attempts. Suicide Life Threat Behav. 2005 Dec;35(6):671-80. doi: 10.1521/suli.2005.35.6.671. PMID 16552982
- [Result] Bauer MS, Wisniewski SR, Marangell LB, Chessick CA, Allen MH, Dennehy EB, Miklowitz DJ, Thase ME, Sachs GS. Are antidepressants associated with new-onset suicidality in bipolar disorder? A prospective study of participants in the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). J Clin Psychiatry. 2006 Jan;67(1):48-55. doi: 10.4088/jcp.v67n0108. PMID 16426088
- [Result] Miklowitz DJ, Wisniewski SR, Miyahara S, Otto MW, Sachs GS. Perceived criticism from family members as a predictor of the one-year course of bipolar disorder. Psychiatry Res. 2005 Sep 15;136(2-3):101-11. doi: 10.1016/j.psychres.2005.04.005. PMID 16023735
- [Result] Perlis RH, Delbello MP, Miyahara S, Wisniewski SR, Sachs GS, Nierenberg AA; STEP-BD investigators. Revisiting depressive-prone bipolar disorder: polarity of initial mood episode and disease course among bipolar I systematic treatment enhancement program for bipolar disorder participants. Biol Psychiatry. 2005 Oct 1;58(7):549-53. doi: 10.1016/j.biopsych.2005.07.029. Epub 2005 Sep 28. PMID 16197928
- [Result] Baldassano CF, Marangell LB, Gyulai L, Ghaemi SN, Joffe H, Kim DR, Sagduyu K, Truman CJ, Wisniewski SR, Sachs GS, Cohen LS. Gender differences in bipolar disorder: retrospective data from the first 500 STEP-BD participants. Bipolar Disord. 2005 Oct;7(5):465-70. doi: 10.1111/j.1399-5618.2005.00237.x. PMID 16176440
- [Result] Mansour HA, Talkowski ME, Wood J, Pless L, Bamne M, Chowdari KV, Allen M, Bowden CL, Calabrese J, El-Mallakh RS, Fagiolini A, Faraone SV, Fossey MD, Friedman ES, Gyulai L, Hauser P, Ketter TA, Loftis JM, Marangell LB, Miklowitz DJ, Nierenberg AA, Patel J, Sachs GS, Sklar P, Smoller JW, Thase ME, Frank E, Kupfer DJ, Nimgaonkar VL. Serotonin gene polymorphisms and bipolar I disorder: focus on the serotonin transporter. Ann Med. 2005;37(8):590-602. doi: 10.1080/07853890500357428. PMID 16338761
- [Result] Ghaemi SN, Hsu DJ, Thase ME, Wisniewski SR, Nierenberg AA, Miyahara S, Sachs G. Pharmacological Treatment Patterns at Study Entry for the First 500 STEP-BD Participants. Psychiatr Serv. 2006 May;57(5):660-5. doi: 10.1176/ps.2006.57.5.660. PMID 16675760
- [Result] Miklowitz DJ, Otto MW, Wisniewski SR, Araga M, Frank E, Reilly-Harrington NA, Lembke A, Sachs GS. Psychotherapy, symptom outcomes, and role functioning over one year among patients with bipolar disorder. Psychiatr Serv. 2006 Jul;57(7):959-65. doi: 10.1176/ps.2006.57.7.959. PMID 16816280
- [Result] Otto MW, Simon NM, Wisniewski SR, Miklowitz DJ, Kogan JN, Reilly-Harrington NA, Frank E, Nierenberg AA, Marangell LB, Sagduyu K, Weiss RD, Miyahara S, Thas ME, Sachs GS, Pollack MH; STEP-BD Investigators. Prospective 12-month course of bipolar disorder in out-patients with and without comorbid anxiety disorders. Br J Psychiatry. 2006 Jul;189:20-5. doi: 10.1192/bjp.bp.104.007773. PMID 16816301
- [Result] Friedman E, Gyulai L, Bhargava M, Landen M, Wisniewski S, Foris J, Ostacher M, Medina R, Thase M. Seasonal changes in clinical status in bipolar disorder: a prospective study in 1000 STEP-BD patients. Acta Psychiatr Scand. 2006 Jun;113(6):510-7. doi: 10.1111/j.1600-0447.2005.00701.x. PMID 16677228
- [Result] Wolff N, Perlick DA, Kaczynski R, Calabrese J, Nierenberg A, Miklowitz DJ. Modeling costs and burden of informal caregiving for persons with bipolar disorder. J Ment Health Policy Econ. 2006 Jun;9(2):99-110. PMID 17007487
- [Result] Marangell LB, Suppes T, Ketter TA, Dennehy EB, Zboyan H, Kertz B, Nierenberg A, Calabrese J, Wisniewski SR, Sachs G. Omega-3 fatty acids in bipolar disorder: clinical and research considerations. Prostaglandins Leukot Essent Fatty Acids. 2006 Oct-Nov;75(4-5):315-21. doi: 10.1016/j.plefa.2006.07.008. Epub 2006 Aug 22. PMID 16928441
- [Result] Marangell LB, Bauer MS, Dennehy EB, Wisniewski SR, Allen MH, Miklowitz DJ, Oquendo MA, Frank E, Perlis RH, Martinez JM, Fagiolini A, Otto MW, Chessick CA, Zboyan HA, Miyahara S, Sachs G, Thase ME. Prospective predictors of suicide and suicide attempts in 1,556 patients with bipolar disorders followed for up to 2 years. Bipolar Disord. 2006 Oct;8(5 Pt 2):566-75. doi: 10.1111/j.1399-5618.2006.00369.x. PMID 17042830
- [Result] Miklowitz DJ, Otto MW. Psychosocial interventions for bipolar disorder: a review of literature and introduction of the systematic treatment enhancement program. Psychopharmacol Bull. 2007;40(4):116-31. PMID 18227782
- [Result] Sachs GS, Nierenberg AA, Calabrese JR, Marangell LB, Wisniewski SR, Gyulai L, Friedman ES, Bowden CL, Fossey MD, Ostacher MJ, Ketter TA, Patel J, Hauser P, Rapport D, Martinez JM, Allen MH, Miklowitz DJ, Otto MW, Dennehy EB, Thase ME. Effectiveness of adjunctive antidepressant treatment for bipolar depression. N Engl J Med. 2007 Apr 26;356(17):1711-22. doi: 10.1056/NEJMoa064135. Epub 2007 Mar 28. PMID 17392295
- [Result] Miklowitz DJ, Otto MW, Frank E, Reilly-Harrington NA, Wisniewski SR, Kogan JN, Nierenberg AA, Calabrese JR, Marangell LB, Gyulai L, Araga M, Gonzalez JM, Shirley ER, Thase ME, Sachs GS. Psychosocial treatments for bipolar depression: a 1-year randomized trial from the Systematic Treatment Enhancement Program. Arch Gen Psychiatry. 2007 Apr;64(4):419-26. doi: 10.1001/archpsyc.64.4.419. PMID 17404119
- [Derived] Prisciandaro JJ, Tolliver BK, DeSantis SM. Identification and initial validation of empirically derived bipolar symptom states from a large longitudinal dataset: an application of hidden Markov modeling to the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) study. Psychol Med. 2019 May;49(7):1102-1108. doi: 10.1017/S0033291718002143. Epub 2018 Aug 29. PMID 30153871
- [Derived] Bareis N, Lu J, Kirkwood CK, Kornstein SG, Wu E, Mezuk B. Identifying clinical net benefit of psychotropic medication use with latent variable techniques: Evidence from Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). J Affect Disord. 2018 Oct 1;238:147-155. doi: 10.1016/j.jad.2018.05.063. Epub 2018 May 29. PMID 29883936
- [Derived] Slyepchenko A, Frey BN, Lafer B, Nierenberg AA, Sachs GS, Dias RS. Increased illness burden in women with comorbid bipolar and premenstrual dysphoric disorder: data from 1 099 women from STEP-BD study. Acta Psychiatr Scand. 2017 Nov;136(5):473-482. doi: 10.1111/acps.12797. Epub 2017 Aug 28. PMID 28846801
- [Derived] Mizushima J, Uchida H, Tada M, Suzuki T, Mimura M, Nio S. Early Improvement of Specific Symptoms Predicts Subsequent Recovery in Bipolar Depression: Reanalysis of the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) Data. J Clin Psychiatry. 2017 Feb;78(2):e146-e151. doi: 10.4088/JCP.15m10573. PMID 28234437
- [Derived] Prisciandaro JJ, Tolliver BK. An item response theory evaluation of the young mania rating scale and the montgomery-asberg depression rating scale in the systematic treatment enhancement program for bipolar disorder (STEP-BD). J Affect Disord. 2016 Nov 15;205:73-80. doi: 10.1016/j.jad.2016.06.062. Epub 2016 Jul 13. PMID 27420134
- [Derived] Ballard ED, Vande Voort JL, Luckenbaugh DA, Machado-Vieira R, Tohen M, Zarate CA. Acute risk factors for suicide attempts and death: prospective findings from the STEP-BD study. Bipolar Disord. 2016 Jun;18(4):363-72. doi: 10.1111/bdi.12397. Epub 2016 May 27. PMID 27233466
- [Derived] Tada M, Uchida H, Mizushima J, Suzuki T, Mimura M, Nio S. Antidepressant dose and treatment response in bipolar depression: Reanalysis of the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) data. J Psychiatr Res. 2015 Sep;68:151-6. doi: 10.1016/j.jpsychires.2015.06.015. Epub 2015 Jun 23. PMID 26228414
- [Derived] Prisciandaro JJ, Tolliver BK. Evidence for the continuous latent structure of mania and depression in out-patients with bipolar disorder: results from the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). Psychol Med. 2015;45(12):2595-603. doi: 10.1017/S0033291715000513. Epub 2015 Apr 17. PMID 25881582
- [Derived] Stange JP, Sylvia LG, da Silva Magalhaes PV, Miklowitz DJ, Otto MW, Frank E, Berk M, Nierenberg AA, Deckersbach T. Extreme attributions predict the course of bipolar depression: results from the STEP-BD randomized controlled trial of psychosocial treatment. J Clin Psychiatry. 2013 Mar;74(3):249-55. doi: 10.4088/JCP.12m08019. PMID 23561230
- [Derived] Magalhaes PV, Kapczinski F, Nierenberg AA, Deckersbach T, Weisinger D, Dodd S, Berk M. Illness burden and medical comorbidity in the Systematic Treatment Enhancement Program for Bipolar Disorder. Acta Psychiatr Scand. 2012 Apr;125(4):303-8. doi: 10.1111/j.1600-0447.2011.01794.x. Epub 2011 Nov 19. PMID 22098628
- [Derived] Ghaemi SN, Ostacher MM, El-Mallakh RS, Borrelli D, Baldassano CF, Kelley ME, Filkowski MM, Hennen J, Sachs GS, Goodwin FK, Baldessarini RJ. Antidepressant discontinuation in bipolar depression: a Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) randomized clinical trial of long-term effectiveness and safety. J Clin Psychiatry. 2010 Apr;71(4):372-80. doi: 10.4088/JCP.08m04909gre. PMID 20409444
- [Derived] Goldberg JF, Brooks JO 3rd, Kurita K, Hoblyn JC, Ghaemi SN, Perlis RH, Miklowitz DJ, Ketter TA, Sachs GS, Thase ME. Depressive illness burden associated with complex polypharmacy in patients with bipolar disorder: findings from the STEP-BD. J Clin Psychiatry. 2009 Feb;70(2):155-62. doi: 10.4088/jcp.08m04301. Epub 2009 Feb 10. PMID 19210946
- [Derived] Nowakowska C, Sachs GS, Zarate CA Jr, Marangell LB, Calabrese JR, Goldberg JF, Ketter TA. Increased rate of non-right-handedness in patients with bipolar disorder. J Clin Psychiatry. 2008 May;69(5):866-7. doi: 10.4088/jcp.v69n0522g. No abstract available. PMID 18681768
- [Derived] Marangell LB, Dennehy EB, Wisniewski SR, Bauer MS, Miyahara S, Allen MH, Martinez M, Al Jurdi RK, Thase ME. Case-control analyses of the impact of pharmacotherapy on prospectively observed suicide attempts and completed suicides in bipolar disorder: findings from STEP-BD. J Clin Psychiatry. 2008 Jun;69(6):916-22. doi: 10.4088/jcp.v69n0605. PMID 18399724
- [Derived] Miklowitz DJ, Otto MW, Frank E, Reilly-Harrington NA, Kogan JN, Sachs GS, Thase ME, Calabrese JR, Marangell LB, Ostacher MJ, Patel J, Thomas MR, Araga M, Gonzalez JM, Wisniewski SR. Intensive psychosocial intervention enhances functioning in patients with bipolar depression: results from a 9-month randomized controlled trial. Am J Psychiatry. 2007 Sep;164(9):1340-7. doi: 10.1176/appi.ajp.2007.07020311. PMID 17728418